CLINICAL TRIAL: NCT03661398
Title: Clinical Investigation of the Caisson Transcatheter Mitral Valve Replacement (TMVR) System for Percutaneous Mitral Valve Replacement in Patients With Symptomatic Mitral Regurgitation
Brief Title: Caisson Transcatheter Mitral Valve Replacement (TMVR)
Acronym: INTERLUDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Caisson Interventional LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT-001
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Mitral Regurgitation; Mitral Valve Disease; Mitral Valve Failure; Mitral Disease; Valve Heart Disease; Valve Disease, Heart
Keywords: Percutaneous mitral valve replacement; Trans-septal mitral valve replacement; Transcatheter mitral valve replacement; TMVR; Primary MR; Secondary MR; Structural Heart Disease; Heart Failure; Degenerative Mitral Valve Disease; Functional Mitral Valve Disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Disease; Heart Valve Diseases; Heart Failure | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcatheter Mitral Valve Replacement (Experimental): Patients with symptomatic mitral regurgitation (garde 3 or 4), determined to be a high risk for cardiovascular surgery, will be treated with the Caisson Transcatheter Mitral Valve Replacement (TMVR) System
  Interventions: Device: Transcatheter Mitral Valve Replacement

INTERVENTIONS:
Device: Transcatheter Mitral Valve Replacement — All eligible patients will be in the treatment arm for treatment with the Caisson Transcatheter Mitral Valve Replacement (TMVR) System. There is no control (comparator) arm for this study.
  Other Names: Caisson Transcatheter Mitral Valve Replacement (TMVR) System

SUMMARY:
The purpose of this study is to assess the safety and performance of Transcatheter Mitral Valve Replacement (TMVR) system for the treatment of severe, symptomatic mitral regurgitation (MR).

DETAILED DESCRIPTION:
The treatment guidelines for valvular heart disease indicate that surgical correction of primary mitral valve regurgitation (MR) is a Class I recommendation. Recent evidence indicates that valve replacement is at least as effective as repair in both primary and secondary MR patients. However, many patients are not referred for surgery as they are considered to be too high of a risk to undergo on-pump, open-heart procedures. Percutaneous aortic valve replacement has made treatment of stenosed aortic valves available to high-risk surgical patients who would have otherwise been medically managed. Percutaneous mitral valve (MV) replacement offers similar advantages. The feasibility of percutaneous MV replacement has been demonstrated in early feasibility studies. To meet this medical need, Caisson Interventional has developed a percutaneous delivery system for a bioprosthetic mitral valve. As with patients with aortic valve (AV) deficiencies, this device can be used to provide needed therapy to patients who might not otherwise receive treatment beyond medical therapy. This study will provide information on the safety and performance of this system.

ELIGIBILITY:
Inclusion Criteria:

* Has severe mitral regurgitation
* New York Heart Association (NYHA) Class II, III, IVa or heart failure
* High risk for cardiovascular surgery

Exclusion Criteria:

* Excessive calcification or thickening of mitral valve annulus
* Severe mitral stenosis, fused commissures, valvular vegetation or mass
* Left ventricular end diastolic dimension > 7cm
* Left ventricular outflow tract obstruction
* Severe right ventricular dysfunction
* Stroke within 90 days; transient ischemic attack or myocardial infarction within 30 days of the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients without Major Adverse Events (MAEs) | 30 days
  Freedom from major adverse events including death, stroke, myocardial infarction and surgical reintervention through 30 days

SECONDARY OUTCOMES:
Number of patients with successful delivery and implantation of the prosthetic valve (technical success) | Intra-operative
  Successful delivery and retrieval of the transcatheter mitral valve delivery system; deployment and correct positioning (via intraoperative imaging) in the appropriate anatomic location of prosthetic valve with no requirement for additional surgery
Number of living, stroke-free patients with prosthetic valve in place (device success) | 30 days
  Patient is alive, stroke-free, original intended device in place (echo), no mitral valve surgical re-intervention required

CONTACTS AND LOCATIONS:
Overall Officials: Mat Williams, M.D., Principal Investigator — NYU Langone Medical Center
Locations (1):
- Pennsylvania State University, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No